CLINICAL TRIAL: NCT04255732
Title: Comparison Between Two Wide-field Imaging Systems on the Extent of Retinal Periphery Area Viewing
Brief Title: Comparison of Wide-field Retinal Imaging
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Prim. Prof. Dr. Oliver Findl, MBA (Other)
Responsible Party: Sponsor-Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Head of Ophthalmology Department, principal investigator, Vienna Institute for Research in Ocular Surgery
Organization: Vienna Institute for Research in Ocular Surgery (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UWF
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2020-10-06 (Actual); Status verified 2020-10

CONDITIONS: Retinal Disease
Keywords: retinal imaging; wide field
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Extent of retinal periphery area viewing (Other): For the 30 patients fundus photography will be performed using two ultra-wide-field imaging systems.
  Interventions: Device: extent of retinal area viewing Optos, Daytona, Optos PLC, Dunfermline, UK; Device: extent of retinal area viewing Clarus, 500 Carl Zeiss, Meditec AG, Jena, Germany

INTERVENTIONS:
Device: extent of retinal area viewing Optos, Daytona, Optos PLC, Dunfermline, UK — Comparison of the extent of retinal periphery view between two wide field imaging devices.
Device: extent of retinal area viewing Clarus, 500 Carl Zeiss, Meditec AG, Jena, Germany — Comparison of the extent of retinal periphery view between two wide field imaging devices.

SUMMARY:
Fundus imaging has become an integral tool in retinal diagnosis. Although single-field fundus photography covers a vital region of the retina, it leaves a large portion of the periphery undiscovered.

Ultra-wide-field imaging systems allowed for visualization of peripheral perfusion abnormalities in myopic eyes that were previously unknown.

In Austria, there are two different wide-field imaging systems available. The first device on the market was the Optos (Optos PLC, Dunfermline, UK) and several years later the Clarus 500 (Carl Zeiss, Meditec AG, Jena, Germany) was introduced.

DETAILED DESCRIPTION:
While both of the studied imaging systems have the possibility of a 200° view of the retina, we would asses if the differences between the two devices affect the extent of retinal periphery view and if ocular ametropies which come with different retinal pathologies would affect the retinal periphery assessment.

Aim: To compare two CE-marked imaging systems concerning the extent of retinal periphery area viewing.

We would like to perform a prospective observational study that would include patients divided into three groups: myopic patients, hyperopic and emmetropic patients.

Fundus photography will be performed using two ultra-wide-field imaging systems (Optos, Daytona, Optos PLC, Dunfermline, UK and Clarus, 500 Carl Zeiss, Meditec AG, Jena, Germany), performed by the same investigator.

All images with sufficient quality will be exported and saved to hard-disk. The difference in periphery view will be investigated as follows: two retinal photos for each patient will be imported into Photoshop CS6 image-editing system (Adobe, version 13.0.0) where the anatomical landmarks will be matched for each image and the borders will be compared to see if there are differences in retinal periphery area viewing between the two devices.

ELIGIBILITY:
Inclusion Criteria:

* Patient over 21 years old
* Myopic (at least -5.00Dsph), hyperopic (over +3.00Dsph) and emmetropic patients
* Written informed consent prior to any study specific action.

Exclusion Criteria:

* Extensive cataract or severe corneal scaring that would affect image quality
* Fixation problems, nystagmus
* pregnancy- for women in reproductive age a pregnancy test will be performed.

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-08-07 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
difference in retinal periphery viewing between the two devices | 7 months
  Extent of retinal periphery area viewing (the difference in periphery area between the two devices). Images of the same patients will be compared to determine the degree of periphery viewing for the two devices.

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, Prof., Principal Investigator — VIROS, Hanusch Hospital Vienna
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No